CLINICAL TRIAL: NCT06940323
Title: Pregnancy Registry, Infants, Serum/Milk Analysis (PRISMA): Pregnancy Registry for Women With Chronic Conditions
Brief Title: Pregnancy Registry, Infants, Serum/Milk Analysis (PRISMA)
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: PRISMA
Record Dates: First submitted 2025-03-19; First posted 2025-04-23 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis; Clinically Isolated Syndrome; NMOSD; Myasthenia Gravis
MeSH Terms: conditions — Multiple Sclerosis; Myasthenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Maternal blood, stool, vaginal microbiome, breastmilk sample, and infant stool sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Healthy Controls: Healthy adult women who are planning pregnancy, currently pregnant, or postpartum.
- Multiple sclerosis (MS): Adult women diagnosed with multiple sclerosis (MS) who are planning pregnancy, currently pregnant, or postpartum.
- Clinically isolated syndrome (CIS): Adult women diagnosed with clinically isolated syndrome (CIS) who are planning pregnancy, currently pregnant, or postpartum.
- Neuromyelitis optica spectrum disorder (NMOSD): Adult women diagnosed with neuromyelitis optica spectrum disorder (NMOSD) who are planning pregnancy, currently pregnant, or postpartum.
- Myasthenia gravis: Adult women diagnosed with myasthenia gravis who are planning pregnancy, currently pregnant, or postpartum.

SUMMARY:
PRISMA, is a pregnancy registry study, focused on comprehensively collecting information about pregnancy in women with chronic neurological conditions from across the United States and internationally.

Depending on their specific condition (MS, CIS, NMOSD, or other) and their specific treatment, participants will be asked to contribute to different aspects of the study. (1) The biosamples will be blood, breast milk, infant stool, maternal stool and vaginal swab samples, collected at specific time points. (2) The online surveys will be collected at specific time points. All study activities will be discussed with participants upon enrollment.

By collecting this information, the investigators hope to gain deeper insights into the relationship between pregnancy, the neurological condition, and maternal and infant health. For example, one of the sub-studies focuses on breast milk collection for women planning postpartum treatment with Ocrevus, Rituxan, Briumvi or Kesimpta.

This study is fully remote and all sample collection is optional, so participants can choose which types of samples they wish to provide. For blood draws, participants can schedule a home visit through ExamOne, making participation even more convenient.

The investigators aim to enroll women with chronic neurological conditions who are planning pregnancy, currently pregnant, or within one year postpartum.

DETAILED DESCRIPTION:
The aim of this project is to develop a repository of samples for women who are pregnant and have chronic conditions, including demyelinating diseases -- either multiple sclerosis (MS), clinically isolated syndrome (CIS) or NMOSD (neuromyelitis optica spectrum disorders), chronic inflammation --- inflammatory bowel disease (IBD), rheumatoid arthritis (RA), lupus, myasthenia gravis (MG), primary headache disorders, or other chronic neurological conditions. Please note that the investigators refer to "MS" in the rest of the application.

This repository will include:

1. Maternal Outcomes (disease-related outcomes, depression, social support, breastfeeding and pregnancy-related outcomes):

   * Obtained via interviews, surveys, and medical record review during pregnancy planning, pregnancy (Baseline and 36w gestation) and postpartum (1, 4, 8, 12M)
   * Maternal radiographic information will be collected from data available in the medical records. [Radiographic information will be information captured from the medical record, not obtained during the study visits. No radiology exams will be conducted as part of this research study. If deemed necessary for the subject's routine clinical care, the investigators will record the results of an MRI within 12M postpartum.]
2. Infant Outcomes (growth, development, immunization, infection, breastfeeding, etc.)

   * Obtained via medical record review (up to 12M)
   * Monitored via maternal completion of the Ages and Stages Questionnaires-Version 3 (ASQ3) to track infant development outcomes (communication, gross motor, fine motor, problem solving, and person-social) at 2, 4, 6, 8, 10, and 12M of age.
3. Biospecimen Collection, Storage & Later Batch Analysis:

   * Maternal blood samples will be collected for up to the following time points: Baseline (including if planning pregnancy), 3M gestation, 6M gestation, 8M gestation, 1M postpartum, 3M postpartum, and 6M postpartum. Samples will be processed and stored as serum, plasma and peripheral blood mononuclear cells (PBMCs).
   * Serial breastmilk samples will be collected, for both before and after treatment if applicable, and up to 2-3 years postpartum. These samples will be used to determine the concentrations of medications in breastmilk relative to maternal serum.
   * Serial maternal and infant gut microbiome samples will be collected before and after treatment (anytime during the lactation period which can extend up to 2-3 years postpartum) to determine the effect of mAb treatment on gut microbial populations in mothers and infants. Mothers will be asked to complete food frequency questionnaires for themselves and their infants at the time of each sample collection.
   * Maternal vaginal swab sample will be collected in their 36 weeks of gestation (OR 8M pregnancy) to determine the effect of mAb treatment on vaginal microbial populations in mothers. Mothers will be asked to complete questionnaires regarding their diet and medication for themselves at the time of each sample collection.
   * Serial maternal blood samples will be collected (including before and post treatment) anytime up to 2-3 years postpartum. These samples will be used to determine concentrations of medications in breastmilk relative to serum and to determine the effect of maternal treatment on mother and infant gut microbiome.

     * Timing of sample collection for participants treated with mAb will depend on the treatment type, dosing and infusion schedule.

Participants who are healthy controls or who are not receiving specific medications of interest will provide

* A single breastmilk sample at 2M, 3M, and 4M
* A maternal and infant gut microbiome sample at 2M, 3M, and 4M postpartum
* Maternal vaginal swab sample at 36 weeks of gestation (OR 8M pregnancy).
* Maternal blood samples will be collected at corresponding timepoints 2M, 3M and 4M postpartum (to be processed and stored as serum, plasma, and PBMCs)

ELIGIBILITY:
Inclusion Criteria:

* Pregnant or contemplating pregnancy
* Female, aged 18 to 64 years
* Diagnosis of one of the following conditions:
* Clinically Isolated Syndrome (CIS) or Multiple Sclerosis (MS), based on the 2010 McDonald Criteria
* Neuromyelitis Optica Spectrum Disorder (NMOSD)
* Inflammatory Bowel Disease (IBD)
* Rheumatoid Arthritis (RA)
* Myasthenia Gravis
* Lupus
* Other chronic neurological conditions
* Willing to provide biosamples and/or complete surveys at specified timepoints
* Women without a chronic condition who are pregnant or contemplating pregnancy (as part of the control group)

Exclusion Criteria:

- Unwillingness to provide informed consent

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult women diagnosed with multiple sclerosis (MS), clinically isolated syndrome (CIS), Neuromyelitis optica spectrum disorder (NMOSD), and/or myasthenia gravis who are planning pregnancy, currently pregnant, or postpartum.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-03-21 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2035-06 (Estimated)

PRIMARY OUTCOMES:
Maternal Disease Activity During Pregnancy and Postpartum Assessed by Expanded Disability Status Scale (EDSS) | From pre-pregnancy (if applicable) through 12 months postpartum
  Changes in maternal disease activity will be assessed using the Expanded Disability Status Scale (EDSS) for individuals with multiple sclerosis (scored from 0 to 10, with higher scores indicating greater disability). Data will be collected via medical record review and participant self-report questionnaires.
Maternal Disease Activity During Pregnancy and Postpartum Assessed by MRI Findings | From pre-pregnancy (if applicable) through 12 months postpartum
  Changes in maternal disease activity will be assessed using magnetic resonance imaging (MRI) findings, including gadolinium-enhancing lesions, new or enlarging T2 lesions, and brain atrophy. Data will be collected via medical record review.
Maternal Disease Treatment Course During Pregnancy and Postpartum Assessed by Disease Modifying Therapy (DMT) Use | From pre-pregnancy (if applicable) through 12 months postpartum
  The maternal disease treatment course will be evaluated through an assessment of Disease Modifying Therapy (DMT) used pre-pregnancy to postpartum. This includes the specific type of DMT used in the pre-pregnancy period, any modifications or discontinuation of therapy during pregnancy, and the resumption or initiation of DMTs in the postpartum period. Data will be obtained through medical record review.
Maternal Disease Activity During Pregnancy and Postpartum Assessed by Clinical Relapse Rates | From pre-pregnancy (if applicable) through 12 months postpartum
  Changes in maternal disease activity will be assessed using the clinical relapse rate. Relapses will be identified based on medical record review and participant self-report questionnaires administered at regular intervals. Additional information, such as the timing, severity, and treatment of relapses, will be collected when available.

SECONDARY OUTCOMES:
Infant Growth and Development Outcomes Assessed by Chart Review and ASQ-3 | From birth through 12 months postpartum
  Infant growth data (weight, length, head circumference) will be extracted from routine clinical records from Well-Child Care Visits up to 12 months. Developmental milestones will be assessed using the Ages and Stages Questionnaire, Version 3 (ASQ-3), administered at 2, 4, 6, 8, 10, and 12 months postpartum. ASQ-3 scores are age-specific and help assess infant communication, motor, problem-solving, and social-emotional development. Higher scores generally indicate better developmental progress.
Detection and Concentration of Monoclonal Antibodies in Breastmilk | From first infusion postpartum through 12 months postpartum
  Breastmilk samples will be collected following postpartum infusions of anti-B cell therapies (e.g., ocrelizumab, rituximab), natalizumab, or monoclonal antibodies targeting calcitonin gene-related peptide (CGRP) or its receptor. Samples will be collected across 6 timepoints around the first postpartum infusion (pre-infusion; 7 days, 20 days, 30 days, 60 days, and 90 days post-infusion). Samples will be analyzed to detect the presence and concentration of these therapies in breastmilk and predict the relative transfer of medication to infants through breastmilk. Information about breastfeeding behavior including whether participants are exclusively breastfeeding, mixed feeding, or using formula, will be self-reported through accompanying survey or collected through chart review.
Concentration of Monoclonal Antibodies and Disease-Related Biomarkers in Maternal Blood | From the planning pregnancy (if applicable) to 6 months postpartum
  Maternal blood samples will be collected at various time points: during the planning stage, at 8 months of pregnancy, and during the postpartum period (1, 2, 4, and 6 months postpartum), depending on the participant's ability and willingness to provide a sample. During the postpartum period, a set of blood samples will also be collected pre-infusion, and at 30 and 60 days post-infusion, either separately or in conjunction with other postpartum time points. These samples will be analyzed to determine serum drug levels for pharmacokinetic evaluation, as well as to assess other biomarkers of interest.
Maternal Fatigue During Pregnancy and Postpartum Assessed by Modified Fatigue Impact Scale (MFIS) | From pre-pregnancy (if applicable) through 12 months postpartum
  Fatigue will be assessed using the Modified Fatigue Impact Scale (MFIS), which evaluates the perceived impact of fatigue on cognitive, physical, and psychosocial functioning. Scores range from 0 to 84. Higher scores indicate greater fatigue impact. This will be administered at baseline, 8 months of pregnancy, and during the postpartum period at 1, 4, 8, and 12 months.
Maternal Sleep Quality During Pregnancy and Postpartum Assessed by Medical Outcomes Study Sleep Scale (MOS-SS) | From pre-pregnancy (if applicable) through 12 months postpartum
  Sleep quality will be measured using the Medical Outcomes Study Sleep Scale (MOS-SS), which evaluates multiple dimensions of sleep such as sleep disturbance, snoring, and sleep adequacy. Scores are standardized, with higher scores generally indicating worse sleep quality, depending on the subscale. The survey will be administered at baseline, 8 months of pregnancy, and during the postpartum period at 1, 4, 8, and 12 months.
Maternal Sleep Quality During Pregnancy and Postpartum Assessed by Epworth-Sleepiness Scale (ESS) | From pre-pregnancy (if applicable) through 12 months postpartum
  Daytime sleepiness will be assessed using the Epworth Sleepiness Scale (ESS), a self-administered questionnaire that measures the general level of daytime sleepiness. The scale includes 8 items with scores ranging from 0 to 24, where higher scores indicate greater daytime sleepiness. The survey will be administered at baseline, 8 months of pregnancy, and during the postpartum period at 1, 4, 8, and 12 months.
Maternal Cognitive Function During Pregnancy and Postpartum Assessed by Multiple Sclerosis Neuropsychological Questionnaire (MSNQ) | From pre-pregnancy (if applicable) through 12 months postpartum
  The Multiple Sclerosis Neuropsychological Questionnaire (MSNQ) will be used to assess cognitive function and neuropsychological symptoms related to multiple sclerosis (MS). This self-reported questionnaire includes multiple domains such as memory, attention, and executive function, to evaluate the cognitive impact of MS during pregnancy and postpartum. Higher scores indicate more cognitive difficulty. This will be administered at baseline, 8 months of pregnancy, and during the postpartum period at 1, 4, 8, and 12 months.
Social Support During Pregnancy and Postpartum Assessed by Medical Outcomes Study Social Support Survey (19-Item Version) | From pre-pregnancy (if applicable) through 12 months postpartum
  The Medical Outcomes Study Social Support Survey (19-Item Version) will assess the level of social support participants feel they have during pregnancy and postpartum. The survey includes items related to emotional, informational, and tangible support. Responses are scored on a 5-point Likert scale, with higher scores indicating greater perceived social support. This will be collected at baseline, 8 months of pregnancy, and during the postpartum period at 1, 4, 8, and 12 months.
Maternal Per-partum Depression Status During Pregnancy and Postpartum Assessed by Hospital Anxiety and Depression Scale (HADS) | From pre-pregnancy (if applicable) through 12 months postpartum
  Maternal mood and depression symptoms will be assessed using the Hospital Anxiety and Depression Scale (HADS), a 14-item scale with subscales for anxiety and depression, each scored from 0 to 21. Higher scores indicate greater symptom severity. The questionnaire will be administered at baseline (pre-pregnancy or early pregnancy), 36 weeks/8 months gestation, and at 1, 4, 8, and 12 months postpartum.
Maternal Per-partum Depression Status During Pregnancy and Postpartum Assessed by Edinburgh Postnatal Depression Scale (EPDS) | From pre-pregnancy (if applicable) through 12 months postpartum
  Maternal mood and depression symptoms will be assessed using the Edinburgh Postnatal Depression Scale (EPDS), a 10-item scale scored from 0 to 30. Higher scores indicate more severe postpartum depression symptoms. The questionnaire will be administered at baseline (pre-pregnancy or early pregnancy), 36 weeks/8 months gestation, and at 1, 4, 8, and 12 months postpartum.
Maternal Per-partum Depression Status During Pregnancy and Postpartum Assessed by Mini International Neuropsychiatric Interview (MINI) | 12 months postpartum
  Maternal mood and depression symptoms will be assessed using Mini International Neuropsychiatric Interview (MINI), a structured diagnostic tool for mental health disorders. The interview includes specific questions and sections designed to assess the presence and severity of depressive symptoms. The questionnaire will be administered through a phone call for a short duration of around 15 minutes at 12 months postpartum.
Maternal Per-partum Depression Status During Pregnancy and Postpartum Assessed by Structured Clinical Interview for DSM-5 (SCID) | 12 months postpartum
  Maternal mood and depression symptoms will be assessed using the Structured Clinical Interview for DSM-5 (SCID), a semi-structured interview to make diagnoses according to the DSM-5 criteria. The questionnaire will be administered at 12 months postpartum by the study clinician.
Maternal Bonding with Infant Assessed by Mother-to-Infant Bonding Scale (MIBS) | From 1 month through 12 months postpartum
  Maternal emotional bonding with the infant will be assessed using the Mother-to-Infant Bonding Scale (MIBS), a self-administered questionnaire designed to screen for potential bonding disorders in the postpartum period. The MIBS consists of 8 items rated on a 4-point Likert scale, with higher scores indicating greater difficulties in mother-infant bonding. The questionnaire will be administered during the postpartum period at 1, 4, 8, and 12 months.
Infant Feeding Practices Assessed by Breastfeeding Questionnaire | From 1 month through 12 months postpartum
  Infant feeding practices will be assessed using a self-administered Breastfeeding Questionnaire, which captures detailed information on breastfeeding initiation, duration, frequency, exclusivity, and supplementation with formula or solid foods. The questionnaire also includes items addressing maternal perceptions, challenges, and reasons for changes in feeding practices. The questionnaire will be administered during the postpartum period at 1, 4, 8, and 12 months.

OTHER OUTCOMES:
Exploratory: Changes in Maternal Gut Microbiome Composition Following Maternal Monoclonal Antibody Treatment | Pre-infusion through 60 days post-infusion
  Stool samples from mothers will be collected at key time points before and after the first maternal monoclonal antibody treatment resumption (pre-infusion; 30 days and 60 days post-infusion) to evaluate changes in gastrointestinal microbial populations.
Exploratory: Changes in Infant Gut Microbiome Composition Following Maternal Monoclonal Antibody Treatment | Pre-infusion through 60 days post-infusion
  Stool samples from infant will be collected at key time points before and after the first maternal monoclonal antibody treatment resumption (pre-infusion; 30 days and 60 days post-infusion) to evaluate changes in gastrointestinal microbial populations.
Exploratory: Infant Medical Problems Inflicting Immune Functions | From delivery through 12 months postpartum
  Immune function of infants whose mothers received anti-B cell therapies, natalizumab, or monoclonal antibodies to calcitonin gene-related peptide (CGRP) or its receptor will be monitored using clinical data (e.g., lymphocyte counts from cord blood and infant bloodwork) when available through standard medical care.
Exploratory: Changes in Maternal Vaginal Microbiome Composition During Pregnancy | 36 weeks of gestation (OR 8M pregnancy)
  Vaginal swab samples from mothers will be collected at a key time point to determine the effect of mAb treatment on vaginal microbial populations in mothers.

CONTACTS AND LOCATIONS:
Overall Officials: Riley Bove, MD, MSc, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California-San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson A, Krysko KM, Rutatangwa A, Krishnakumar T, Chen C, Rowles W, Zhao C, Houtchens MK, Bove R. Clinical and Radiologic Disease Activity in Pregnancy and Postpartum in MS. Neurol Neuroimmunol Neuroinflamm. 2021 Feb 19;8(2):e959. doi: 10.1212/NXI.0000000000000959. Print 2021 Mar. PMID 33608303
- [Background] LaHue SC, Anderson A, Krysko KM, Rutatangwa A, Dorsey MJ, Hale T, Mahadevan U, Rogers EE, Rosenstein MG, Bove R. Transfer of monoclonal antibodies into breastmilk in neurologic and non-neurologic diseases. Neurol Neuroimmunol Neuroinflamm. 2020 May 27;7(4):e769. doi: 10.1212/NXI.0000000000000769. Print 2020 Jul. PMID 32461351
- [Result] Anderson A, Rowles W, Poole S, Balan A, Bevan C, Brandstadter R, Ciplea AI, Cooper J, Fabian M, Hale TW, Jacobs D, Kakara M, Krysko KM, Longbrake EE, Marcus J, Repovic P, Riley CS, Romeo AR, Rutatangwa A, West T, Hellwig K, LaHue SC, Bove R. Anti-CD20 monoclonal antibody therapy in postpartum women with neurological conditions. Ann Clin Transl Neurol. 2023 Nov;10(11):2053-2064. doi: 10.1002/acn3.51893. Epub 2023 Sep 7. PMID 37675826